CLINICAL TRIAL: NCT05426499
Title: Translational PKPD Modeling of Anti-infective Drugs in Children Treated in Pediatric Units on the Example of Selected Antibiotics and Antifungals.
Brief Title: Translational PKPD Modeling of Anti-infective Drugs Used in Pediatric Units.
Status: Recruiting | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Collaborators: University at Buffalo (Other); The Greater Poland Cancer Centre (Other)
Responsible Party: Principal Investigator, Agnieszka Bienert, Full Professor, Poznan University of Medical Sciences
Other Study IDs: 820/21
Record Dates: First submitted 2021-12-17; First posted 2022-06-22 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2024-06

CONDITIONS: Population Modeling of Anti-infective Drugs
Keywords: Population modeling; Pediatric Units; Pharmacokinetics; Pharmacodynamics; Anti-infective drugs; Cefotaxime; Meropeneme; Fluconazole; Isavuconazole; Anidulafingin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Patients requiring cefotaxime treatment: The treatment choice and the recommended dosage will depend on the isolated pathogen. Therapy will be based on the SmPC of the appropriate drug.
  Interventions: Drug: Patients requiring cefotaxime treatment
- Patients requiring meropenem treatment: The treatment choice and the recommended dosage will depend on the isolated pathogen. Therapy will be based on the SmPC of the appropriate drug.
  Interventions: Drug: Patients requiring meropenem treatment
- Patients requiring fluconazole treatment: The treatment choice and the recommended dosage will depend on the isolated pathogen. Therapy will be based on the SmPC of the appropriate drug.
  Interventions: Drug: Patients requiring fluconazole treatment
- Patients requiring isavuconazole treatment: The treatment choice and the recommended dosage will depend on the isolated pathogen. Therapy will be based on the SmPC of the appropriate drug.
  Interventions: Drug: Patients requiring isavuconazole treatment
- Patients requiring anidulafungin treatment: The treatment choice and the recommended dosage will depend on the isolated pathogen. Therapy will be based on the SmPC of the appropriate drug.
  Interventions: Drug: Patients requiring anidulafungin treatment

INTERVENTIONS:
Drug: Patients requiring cefotaxime treatment — Dosage according to SmPC
  Groups: Patients requiring cefotaxime treatment
Drug: Patients requiring meropenem treatment — Dosage according to SmPC
  Groups: Patients requiring meropenem treatment
Drug: Patients requiring fluconazole treatment — Dosage according to SmPC
  Groups: Patients requiring fluconazole treatment
Drug: Patients requiring isavuconazole treatment — Dosage according to SmPC
  Groups: Patients requiring isavuconazole treatment
Drug: Patients requiring anidulafungin treatment — Dosage according to SmPC
  Groups: Patients requiring anidulafungin treatment

SUMMARY:
Pharmacokinetic and pharmacodynamic modeling (PKPD) is becoming an essential tool for optimizing pharmacotherapy. Building mechanistic models allows determining the relationship between the dose, concentration, pharmacological effect, and side effects in various populations. The growing resistance to drugs among bacteria is a challenge for medicine, and the progress in pharmacometrics enables us to make rational clinical decisions. A particular group of patients is children with differences in PK and PD of drugs. The lack of clinical studies often forces to extrapolate dosing based on the results obtained in adults. In intensive care units, up to 70-90% of drugs in children are used off-label. Drug agencies point to the importance of the population-based approach to data analysis, especially in infants and children. Under the project, work will focus on the PK and PD of antifungal drugs (fluconazole, isavuconazole, and anidulafungin) and antibiotics (cefotaxime and meropenem) in the pediatric and adult populations. The choice of topic is dictated by the growing need to create PKPD models of the drugs mentioned above in children. The hypothesis is the assumption that using a mathematical model will enable to describe the time course of the drug in the organism, the relationship between the effect and the dose of the medicine and its concentration in the plasma, and the influence of individual factors on the PKPD profile of a drug.

DETAILED DESCRIPTION:
Cefotaxime and meropenem are broad-spectrum antibiotics, most commonly prescribed in pediatric and adult intensive care units. Unfortunately, the applied dosing regimens based on the results obtained in adults or only on drug pharmacokinetics (without taking into account the pharmacodynamic profile) often fail. The situation is additionally complicated by the observed clinically significant drug interactions. The results of published studies indicate the need to develop PKPD models for these drugs in the pediatric and adult populations. Fluconazole, isavuconazole and anidulafungin are the azole anti-fungal drugs and echinocandin. Despite the optimistic results of studies in adults, showing high efficacy, a favorable PK profile, and the safety profile of these therapeutics, there are no studies in children.

The research will be conducted at the Pediatric Clinical Hospital of K. Jonscher, The Greater Poland Cancer Center, and Heliodor Święcicki Clinical Hospital of the Medical University in Poznań. With the approval of the Bioethics Committee, about 150 children and adults will be included in the study. Blood samples will be collected at appropriate time points to investigate the PK profile. The measured pharmacological effect will be the minimum inhibitory concentration (MIC). PKPD indices will be included in the model, depending on the tested drug: T> MIC, Cmax / MIC, and AUC / MIC. The values of covariates that may affect drug PK and PD will be reported. The analysis will consider the polymorphisms of the OAT3 organic anion transporter genes and the MRP4 transport protein. HPLC will examine plasma drug concentration levels in conjunction with UV detection. The Xevo TQ-S micro triple quadrupole mass spectrometer, coupled with ultra-efficient liquid chromatography with the PDA acquity UPLC detector I-class PDA Waters. The genetic polymorphism of selected genes will be tested by real-time PCR using the LightCycler® 480 II Instrument. The PKPD population analysis will be performed by nonlinear modeling of mixed-effects using NONMEM version 7.2.0, the GNU Fortran 9.0 compiler, and Wings for NONMEM and RStudio. The collected data will be used to build hypothetical models using neural networks.

The expected result of the project's primary goal is to build PKPD models of fluconazole, isavuconazole, anidulafungin, cefotaxime, and meropenem in the pediatric and adult populations. According to the final model's principles, they will be evaluated and can serve as a specialized tool for personalizing pharmacotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Obtaining informed consent from the patient/parent of the patient
* A bacterial and fungal infection that requires the use of at least one of the drugs listed based on clinical indications and the attending physician's decision.

Exclusion Criteria:

* Proven allergic reaction to medications used
* No written consent
* Contraindications in SmPC
* Combination therapy with at least two antibacterial drugs and/or at least two antifungal drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients with bacterial and/or fungal infections demanding treatment by cefotaxime, meropenem, fluconazole, isavuconazole, or anidulafungin.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Cefotaxime plasma concentration [ng/ml] | Just before the next dose and at 0.33; 0.66; 1; 2; 4; 6; 8 hours after the start of drug administration
  Measurements of cefotaxime plasma concentrations [ng/ml] before and after dosage of a drug. Blood samples were collected according to the study protocol.
Meropenem plasma concentration [ng/ml] | Just before the next dose and at 1,5; 3; 6; 8 hours after the start of drug administration
  Measurements of meropenem plasma concentrations [ng/ml] before and after dosage of a drug. Blood samples were collected according to the study protocol.
Fluconazole plasma concentration [ng/ml] | Just before the next dose and at 0,5; 1; 3; 10; 24 hours after the start of drug administration
  Measurements of fluconazole plasma concentrations [ng/ml] before and after dosage of a drug. Blood samples were collected according to the study protocol.
Isavuconazole plasma concentration [ng/ml] | Just before the next dose and at 0,25; 0,5; 0,75; 1; 1,25; 1,5; 2; 3; 4; 6; 8; 10; 12; 14; 16; 24 hours after the start of drug administration
  Measurements of isavuconazole plasma concentrations [ng/ml] before and after dosage of a drug. Blood samples were collected according to the study protocol.
Anidulafungin plasma concentration [ng/ml] | Just before the next dose and at 0,5; 1; 1,5; 2; 4; 6; 8; 10; 12; 24 hours after the start of drug administration
  Measurements of anidulafungin plasma concentrations [ng/ml] before and after dosage of a drug. Blood samples were collected according to the study protocol.

SECONDARY OUTCOMES:
Minimum inhibitory concentration | On the first day after patient inclusion.
  The lowest concentration (in μg/mL) of an antibiotic that inhibits the growth of a given strain of bacteria.
Plasma creatinine concentration | On the first and sixth day after patient inclusion.
  Measurement of creatinine concentrations in blood and urine.
Creatinine clearance (CrCl) | On the first and sixth day after patient inclusion.
  Calculation of creatinine clearance (CrCl) based on measurement of creatinine concentration.
Estimated GFR (eGFR) | On the first and sixth day after patient inclusion.
  Calculation of estimated GFR (eGFR) based on measurement of creatinine concentration.
Bilirubin concentration | On the first and sixth day after patient inclusion.
  Measurement of bilirubin concentration
Albumin concentration | On the first and sixth day after patient inclusion.
  Measurement of albumin concentration
AST concentration | On the first and sixth day after patient inclusion.
  Measurement of AST concentration
ALT concentration | On the first and sixth day after patient inclusion.
  Measurement of ALT concentration
GGT concentration | On the first and sixth day after patient inclusion.
  Measurement of GGT concentration
ALP concentration | On the first and sixth day after patient inclusion.
  Measurement of ALP concentration

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Bienert, MSC,PhD, Principal Investigator — Poznań University of Medical Sciences; Alicja Bartkowska-Śniatkowska, MD, PhD, Principal Investigator — Poznań University of Medical Sciences; Edmund Grześkowiak, MSC, PhD, Study Director — Poznań University of Medical Sciences; William J. Jusko, PhD, Study Chair — School of Pharmacy and Pharmaceutical Sciences, Department of Pharmaceutical Sciences
Locations (4):
- Poland (4):
  - Szpital Kliniczny im. Karola Jonschera Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan, Greater Poland Voivodeship
  - Poznan University of Medical Sciences, Department of Clinical Pharmacy and Biopharmacy, Poznan, Greater Poland Voivodeship
  - Szpital Kliniczny im. Heliodora Święcickiego UMP, Poznan, Greater Poland Voivodeship
  - Wielkopolskie Centrum Onkologii, Poznan, Greater Poland Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Pharmacokinetic and pharmacodynamic data (concentration/effect/time profiles) or individuals will be availabla
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available in 6-12 months and available for 5 years
Access Criteria: Scientists